CLINICAL TRIAL: NCT04097652
Title: The Safety and Tolerability After Intravenous Infusion of UMC119-06 in Subjects With Acute Ischemic Stroke.
Brief Title: Mesenchymal Stem Cells for The Treatment of Acute Ischemic Stroke
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meridigen Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMC119-06-01
Record Dates: First submitted 2019-09-17; First posted 2019-09-20 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2022-12

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- UMC119-06 (Experimental): Human Umbilical Cord Derived-Mesenchymal Stem Cells, Single treatment by intravenous infusion.
  Interventions: Biological: UMC119-06

INTERVENTIONS:
Biological: UMC119-06 — Cohort 1: Low does of UMC119-06；Cohort 2: Medium does of UMC119- 06；Cohort 3: High does of UMC119-06

SUMMARY:
The clinical study with UMC119-06 is designed to investigate the safety in patients with acute ischemic stroke ("AIS"). This will be a dose escalation, open-label, single-center study in adult with acute ischemic stroke. UMC119-06 is ex vivo cultured human umbilical cord tissue-derived mensenchymal stem cells product which is intended for treatment of acute ischemic stroke.

DETAILED DESCRIPTION:
Stroke is the second most important cause of mortality and morbidity in the world. Currently, the standard treatment for ischemic stroke is an intravenous tissue plasminogen activator(tPA; alteplase) and/or endovascular thrombectomy. However, the therapeutic time window for these treatments is narrow. Besides, endovascular thrombectomy requires specialized stroke expertise and endovascular skills. Less than 5% of ischemic stroke patients are treated by these therapy and not all patients achieve good outcomes. There is still a lack of therapy for the reduction disability from stroke. In 2018, at least 40 clinical trials intent to treat ischemic stroke using cell therapy. In particular, MSCs have shown great potential in the reduction disability from acute ischemic stroke (AIS). Meridigen is developing UMC119-06, a mesenchymal stem cell derived from human umbilical cord for the treatment of AIS disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of age between ≥ 20 through ≤ 80 years.
2. Subjects who had an onset of ischemic stroke within 48 to 168 hours before start of treatment.
3. Subjects with occurrence of an ischemic stroke with clear motor or speech deficit documented by National Institutes of Health Stroke Scale (NIHSS) score of 5 to 20 (at the baseline assessment) that did not change by ≥4 points from the screening to the baseline assessment.
4. Subjects who had an onset of ischemic stroke with large-artery atherosclerosis or cardioembolism.
5. Subjects with confirmation of hemispheric cortical infarct with brain magnetic resonance imaging (MRI) including diffusion-weighted imaging demonstrating an acute lesion measuring <100 mL.
6. Subjects modified Rankin score of 0 or 1, reported by subject or family, prior to the onset of symptoms of the current stroke.
7. Subjects with body weight of 50 to 90 kgs.
8. Subject or legal guardian is willing to provide written informed consent to participate in the study after reading the informed consent form and the information provided, and has had the opportunity to discuss the study with the investigator or designee.
9. Women of child-bearing potential should have a negative urine pregnancy test prior to administration of investigational product, UNLESS they meet the following criteria:

(1) Post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum Follicle Stimulating Hormone (FSH) levels > 40mIU/mL, OR; (2) 6 weeks post-surgical bilateral oophorectomy with or without hysterectomy

Exclusion Criteria:

1. Subjects with occurrence of a hemorrhagic transformation of ischemic stroke as evidenced by computerized tomography.
2. Subjects with a lacunar a lesion of ≤ 1.5 cm of longest diameter or a brainstem infarct on MRI as the etiology of current stroke symptoms.
3. Subjects with reduced level of consciousness (score of 3 for item 1a of NIHSS).
4. Subjects who experienced seizures since the onset of ischemic stroke.
5. Subjects with significant head trauma (GCS=3~8) or prior stroke within previous 3 months (except transient ischemic attack (TIA)).
6. Subjects with uncontrolled hypertension despite antihypertensive treatments (persistent systolic blood pressure >180 mm Hg or diastolic >110 mm Hg).
7. Subjects with blood glucose concentration <50 mg/dL or >400 mg/dL.
8. Subjects with uncorrected coagulopathy including, but not limited to:

   1. International normalized ratio (INR) >1.4; or
   2. Activated partial thromboplastin time (aPTT) < 28sec or > 50sec ; or
   3. Platelet (PLT) count <100,000/ mm3 or > 700,000/ mm3.
9. Subjects with history of any type of malignancy.
10. Subjects with major surgery (body organs that require anesthesia, such as tumor removal, open chest, heart surgery, abdominal surgery, intracranial surgery, or normal surgery for more than 3 hours, etc.) within previous 30 days.
11. Subjects who are pregnant (or plan to become pregnant within 3 months of investigational product treatment) or lactating.
12. Subjects who have a significant illness as judged by principal investigator (PI) including, but not limited to:

    1. Severe kidney disease requiring hemodialysis or peritoneal dialysis; or
    2. Advanced liver disease such as liver cirrhosis; or
    3. Severe congestive heart failure (NYHA class 3 and 4); or
    4. Severe pulmonary dysfunction, including severe chronic obstructive pulmonary disease (COPD) and history of lung resection; or
    5. A known history of alcohol abuse or drug abuse within the 6 months before study drug administration, or a history of substance abuse deemed significant by the investigator; or
    6. A known history of severe allergic such as anaphylactic reactions; or
    7. A known history of allergy or hypersensitivity to any component of the formulation (normal saline and human serum albumin); or
    8. A known history of Alzheimer's disease or other dementias, Parkinson's disease, or any other neurological disorder that in the opinion of the trial doctor would affect their ability to participate in the trial or confound study assessments;
13. Subjects who have the following conditions in laboratory tests;

    1. >2 × upper limit of normal (ULN) for alanine aminotransferase (ALT) or aspartate aminotransferase (AST); or
    2. >2 × ULN for serum creatinine;
14. Subjects who are known to be infected with HIV.
15. Subjects who cannot have CT or MRI test.
16. Subjects unable to return for follow-up visits for clinical evaluation, laboratory studies, or imaging evaluation.
17. Subjects who participated in another clinical study of new investigational therapies or has received an investigational therapy within 1 year before the study drug administration.
18. Subjects who have the following medical history including:

    1. Autoimmune disease such as anti-phospholipid syndrome.
    2. Protein C deficiency.
    3. Protein S deficiency.
    4. Sickle cell anemia.
    5. Deep vein thrombosis.
    6. Pulmonary embolism
    7. Long-term use of oral contraceptive drug(defined as using oral contraceptive drug continuously more than 30 days)
    8. Controlled drug abuse.
    9. Brain vascular malformations such as moyamoya disease.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2019-12-05 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence and frequency of adverse events related to administration of UMC119-06. | 3 months from the day of administration
  * Incidence of Treatment-Emergent Adverse Events (TEAEs).
  * Incidence of withdrawals due to AEs.

SECONDARY OUTCOMES:
Changes in Modified Rankin Score (mRS) | 15 months from the day of administration
  Improvement in clinical function as assessed by change in Modified Rankin Score (mRS)
Changes in National Institute of Health Stroke Scale (NIHSS) | 15 months from the day of administration
  Improvement in clinical function as assessed by change in National Institute of Health Stroke Scale (NIHSS)
Changes in Barthel Index (BI) | 15 months from the day of administration
  Improvement in clinical function as assessed by change in Barthel Index (BI)
Changes in Brain MRI | 15 months from the day of administration
  Improvement in clinical function as assessed by change in Brain MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University - Shuang Ho Hospital, Ministry of Health and Welfare., New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No